CLINICAL TRIAL: NCT06057233
Title: Quantitative MRI and GABA Spectroscopy to Localize the Epileptic Zone
Brief Title: Innovative MRI to Localize the Epileptic Zone
Acronym: EPI-CATCHER
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: University Grenoble Alps (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 38RC22.0265_EPI-CATCHER; ANR-21-CE17-0031 (Other Grant/Funding Number: ANR); 2022-A01949-34 (Other: IDRCB)
Record Dates: First submitted 2023-09-19; First posted 2023-09-28 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Epilepsy, Temporal Lobe
Keywords: MRI; Quantitative; GABA; MRS
MeSH Terms: conditions — Epilepsy, Temporal Lobe

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Brain resected tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: mqMRI and GABA-MRS data will be collected in patients suffering from mesial temporal lobe epilepsy
  Interventions: Diagnostic Test: mqMRI and GABA-MRS
- Volunteers: mqMRI and GABA-MRS data will be collected in healthy volunteers
  Interventions: Diagnostic Test: mqMRI and GABA-MRS

INTERVENTIONS:
Diagnostic Test: mqMRI and GABA-MRS — multiparametric quantitative MRI (mqMRI) and of GABA-edited magnetic resonance spectroscopy (GABA-MRS)

SUMMARY:
The goal of EPI-CATCHER is to outline the clinical potential of multiparametric quantitative MRI (mqMRI) and of GABA-edited magnetic resonance spectroscopy (GABA-MRS), combined with machine learning tools, as imaging biomarkers to localize and delineate the EZ.

DETAILED DESCRIPTION:
After informed consent, patient candidate to resection surgery will undergo two extra MRI sessions before surgery: one for multiparametric quantitative MRI (mqMRI) and one for GABA-edited magnetic resonance spectroscopy (GABA-MRS) In parallel, a group of healthy volunteers will also undergo the two MRI sessions described above, to collect reference data.

ELIGIBILITY:
Inclusion Criteria:

* Patient group

  * Patients aged 18-65 years,
  * Patients with drug-resistant focal epilepsy,
  * Patients with MTLE suspicion, with normal MRI or hippocampal sclerosis, and candidate for surgery,
  * Negative pregnancy test for child-bearing aged woman,
  * Obtained signed informed consent from patient
* Reference group

  * Male or female, 18-65 years,
  * Obtained signed informed consent from participants,
  * Negative pregnancy test for child-bearing aged woman

Exclusion Criteria:

* Patient group

  * Patient without social security system
  * Inability or unwillingness of the individual to provide written informed consent, according to national regulations.
  * Impossibility of collecting information on exposure (subjects recently arrived in France, foreign language, etc.),
  * Contraindication for MRI,
  * Contraindication for injection of MRI contrast agent (Gd-Chelate),
  * Evidence on neuroimaging (CT or MRI) of a brain lesion in the same hemisphere as the EZ (tumor, stroke, cerebral edema with midline shift and a clinically significant compression of ventricles, or subarachnoid hemorrhage, or intracerebral parenchymal hematoma (petechial small hemorrhages are NOT a non-inclusion criteria),
  * Severe leucoariosis
  * Pre-existing dementia
  * Pregnant, breastfeeding women
* Reference group

  * Person who is participating in another therapeutic trial
  * Person with a psychiatric disorder, an epilepsy, or a brain lesion susceptible to impact the MRI readouts
  * Person without social security system,
  * Inability or unwillingness of the individual to provide written informed consent, according to national regulations,
  * Impossibility of collecting information on exposure (subjects recently arrived in France, foreign language, etc.),
  * Contraindication for MRI
  * Contraindication for injection of MRI contrast agent (Gd-Chelate)
  * Pregnant, breastfeeding woman.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1 : patients with MTLE epilepsy, candidate to resection surgery Group 2 : healthy volunteers, to obtain reference mqMRI and GABA-MRS values
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
EZmri vs EZsdt | 5 years
  The correlation coefficient between the Dice similarity coefficient (= 2 * the Area of Overlap between EZMRI and EZsdt divided by the total number of pixels in EZMRI and EZsdt) and the reduction in seizure frequency (= seizure frequency one year after surgery / seizure frequency at inclusion).

SECONDARY OUTCOMES:
mqMRI : T1 (ms) | 5 years
  Compare, for each patient, the mqMRI parameter values measured in the EZsdt with the mean mqMRI parameter values obtained in the same region across the healthy volunteers
mqMRI : T2 (ms) | 5 years
  Compare, for each patient, the mqMRI parameter values measured in the EZsdt with the mean mqMRI parameter values obtained in the same region across the healthy volunteers
mqMRI : Mean Diffusivity (s/mm²) | 5 years
  Compare, for each patient, the mqMRI parameter values measured in the EZsdt with the mean mqMRI parameter values obtained in the same region across the healthy volunteers
mqMRI : Cerebral Blood Volume (%) | 5 years
  Compare, for each patient, the mqMRI parameter values measured in the EZsdt with the mean mqMRI parameter values obtained in the same region across the healthy volunteers
mqMRI : Blood-Brain Barrier Permeability (%) | 5 years
  Compare, for each patient, the mqMRI parameter values measured in the EZsdt with the mean mqMRI parameter values obtained in the same region across the healthy volunteers
GABA | 5 years
  Compare, for each patient, the amplitude of GABA and other metabolites available using proton MRS (N-acetyl aspartate and N-acetyl-aspartyl-glutamate (NAA) Creatine and phosphocreatine (Cr), Choline (Cho), Myo-inositol, myo-inositol-monophosphate and glycine (mI), Glutamine (Gln), glutamate (Glu), Lipids (LipX), Lactate (Lac)) in the EZsdt with the mean values obtained in the same region across the healthy volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Kahane, MD, PhD, Principal Investigator — University Grenoble Alps

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boux F, Forbes F, Collomb N, Zub E, Maziere L, de Bock F, Blaquiere M, Stupar V, Depaulis A, Marchi N, Barbier EL. Neurovascular multiparametric MRI defines epileptogenic and seizure propagation regions in experimental mesiotemporal lobe epilepsy. Epilepsia. 2021 May;62(5):1244-1255. doi: 10.1111/epi.16886. Epub 2021 Apr 5. PMID 33818790
- [Background] Hamelin S, Stupar V, Maziere L, Guo J, Labriji W, Liu C, Bretagnolle L, Parrot S, Barbier EL, Depaulis A, Fauvelle F. In vivo gamma-aminobutyric acid increase as a biomarker of the epileptogenic zone: An unbiased metabolomics approach. Epilepsia. 2021 Jan;62(1):163-175. doi: 10.1111/epi.16768. Epub 2020 Dec 1. PMID 33258489